CLINICAL TRIAL: NCT05810103
Title: A Multi-center, Single-arm, Phase І Study of DP303c in Patients With HER2-positive Advanced Solid Tumors
Brief Title: A Study of DP303c in Patients With HER2-positive Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1501-008
Record Dates: First submitted 2023-03-14; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: HER2-positive Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DP303c (Experimental): Eligible patients will be treated with DP303c at 3.0 mg/kg every 3 weeks.
  Interventions: Drug: DP303c

INTERVENTIONS:
Drug: DP303c — DP303c injection, 3.0 mg/kg, every 3 weeks.

SUMMARY:
This is a study of DP303c in patients with HER2-positive advanced solid tumors.

DETAILED DESCRIPTION:
This is a multi-center, single-arm Phase I study to evaluate the pharmacokinetic profile, safety, and initial efficacy of DP303c in patients with HER2-positive advanced solid tumors. Patients will be treated with DP303c injection at 3.0 mg/kg every 3 weeks. Patients will receive DP303c until disease progression, intolerable toxicity, withdrawal of informed consent, death, or any other reasons for treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent;
* Age ≥ 18 years and older;
* Patients with advanced solid tumors confirmed by histology or cytology;
* Received at least 1 line of systemic anti-HER2 therapy or refused systemic therapy for advanced disease states;
* Confirmed to be HER2 positive by local lab;
* The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Life expectancy ≥ 3 months;
* Adequate functions of major organs;
* Female and male patient of childbearing age must agree to take adequate contraceptive measures during the entire study period and through at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Has not recovered from adverse reactions caused by previous anti-tumor treatments to ≤ grade 1 or baseline (refer to NCI CTCAE 5.0) (except for adverse reaction judged by investigators such as alopecia, laboratory tests, etc.);
* History of LVEF < 40%, symptomatic congestive heart failure (CHF), or associated toxicity leading to permanent discontinuation during previous anti-HER2 treatments;
* History of allergy or delayed allergic reaction to any component of study drug that is considered by the investigator to be more severe;
* History of interstitial pneumonia/lung disease requiring steroid treatment;
* The cumulative amount of previous exposure to anthracyclines has reached the certain dosage;
* Treated with strong CYP3A inhibitors or strong CYP3A inducers within 14 days before the first dose of study drug or the presence of concurrent diseases requiring treatment with potent inhibitors or inducers of CYP3A4 during the study treatment;
* History of severe corneal ophthalmopathy;
* Peripheral neuropathy ≥ grade 3 (refer to NCI CTCAE 5.0);
* Symptomatic and unstable cerebral parenchymal metastasis, spinal cord metastasis or compression, and cancerous meningitis;
* Serious or uncontrolled cardiovascular disease;
* Severe chronic or active infection (including tuberculosis infection, etc.) requiring systemic antimicrobial, antifungal, or antiviral therapy within 14 days prior to randomization;
* Active hepatitis B or C;
* History of immunodeficiency diseases, including human immunodeficiency virus (HIV) positive;
* Other circumstances that may interfere with the patient's participation in the study procedures or are inconsistent with the best benefit of the patient's participation or affect the study results: such as a history of severe psychosis, drug or substance abuse, any other clinically important illness or condition, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-03-23 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Day 1,2,3,8, and 15 of cycle 1 and 3, and day 1 of each following cycle (each cycle is 21 days)
Area Under Curve from 0 to the last point (AUC0-last) | Day 1,2,3,8, and 15 of cycle 1 and 3, and day 1 of each following cycle (each cycle is 21 days)
Area Under Curve from t 0 to the infinity (AUC0-inf) | Day 1,2,3,8, and 15 of cycle 1 and 3, and day 1 of each following cycle (each cycle is 21 days)
Time to Reach Peak Serum Concentration (Tmax) | Day 1,2,3,8, and 15 of cycle 1 and 3, and day 1 of each following cycle (each cycle is 21 days)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 12 months
Objective Response Rate (ORR) | Up to approximately 12 months
Duration of Response (DoR) | Up to approximately 12 months
Disease control rate (DCR) | Up to approximately 12 months
Incidence of anti-drug antibodies (ADA) | Day 1, 8, and 15 of cycle 1, and day 1 of each following cycle (each cycle is 21 days)
Incidence of Neutralizing antibodies (Nab) | Day 1, 8, and 15 of cycle 1, and day 1 of each following cycle (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No